CLINICAL TRIAL: NCT05375552
Title: The Effect of Transcranial Direct Current Stimulation Upon Sleep Spindles in Healthy Older Adults: a Pilot Randomised Controlled Study
Brief Title: The Effect of Transcranial Direct Current Stimulation Upon Sleep Spindles in Healthy Older Adults
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has been suspended due to a lack of available staff.
Sponsor: Northumbria University (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NCSR422
Record Dates: First submitted 2022-05-05; First posted 2022-05-16 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Sleep; Aging; Healthy Aging
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transcranial direct current stimulation (Active Comparator): Active transcranial direct current stimulation
  Interventions: Device: Transcranial direct current stimulation
- Placebo transcranial direct current stimulation (Placebo Comparator): Placebo transcranial direct current stimulation
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Participants will experience two repeated 20 minute sessions of tDCS (1.2 mA), with a 10-minute break.

SUMMARY:
A good quantity, and quality, of sleep is crucial for well-being. Evidence strongly indicates that poor sleep quality and quantity is causally involved in the development of dementia; therefore, techniques which can improve sleep in older adults are very likely to prevent or slow down the disease process in dementia.

This project aims to manipulate a specific aspect of sleep in healthy older adults. This: 1) has the potential to prevent the pre-dementia stage of mild cognitive impairment in healthy older adults, and 2) has a direct clinical application to dementia. The overall aim of this project is to investigate if a non-invasive brain stimulation technique called transcranial direct current stimulation (tDCS) can enhance specific brain activity patterns during overnight sleep in healthy older adults.

These brain activity patterns during sleep (called 'sleep spindles') are mechanistically linked to both the physiological restorative and the cognitive function of sleep. Sleep spindles can only be assessed by measuring overnight brain activity during sleep. Sleep spindles are very strongly associated with attention, and memory performance, which are severely affected by dementia. A decrease in sleep spindles is associated with cognitive decline, and predict dementia development. Therefore, enhancing sleep spindle activity in sleep is likely to boost cognition.

Whilst previous research studies have demonstrated that in a sleep laboratory environment, tDCS can manipulate sleep spindles when individuals are in a specific brain state in a nap situation, we are specifically interested in testing tDCS in a home environment. This is because the use of tDCS in a home environment has have a number of advantages over sleep laboratory studies. Specifically, by conducting this study in a home environment, this will maximise the inclusivity of studies involving older adults, and DLB patients, since they will not be required to travel to a sleep laboratory to participate in studies.

The aim of this proof-of-principle study is to investigate if tDCS can manipulate sleep spindles in healthy older adults. It is expected that relative to a placebo stimulation, active stimulation (which exerts an effect upon the brain) will increase sleep spindle activity in healthy older adults.

ELIGIBILITY:
Inclusion Criteria:

• Healthy sleeper older adults aged ≥ 60 years

Exclusion Criteria:

* The presence of self-reported neurodegenerative dementia or other neurological disorders
* Self-reported relevant sleep disorders or disturbances
* Relevant skin allergies
* Concurrent major psychiatric illness
* Significant/severe physical illness or comorbidities
* Metallic or electronic implants

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Slow sleep spindle density | During night immediately after tDCS administration
  PSG-measured slow (11.99Hz) sleep spindle density
Slow sleep spindle amplitude | During night immediately after tDCS administration
  PSG-measured slow (11.99Hz) sleep spindle amplitude.
Fast sleep spindle density | During night immediately after tDCS administration
  PSG-measured fast (13-14.99Hz) sleep spindle density.
Fast sleep spindle amplitude | During night immediately after tDCS administration
  PSG-measured fast (13-14.99Hz) sleep spindle amplitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study will be available from the principal investigator upon reasonable request (after a period of exclusive use (12 months). Our intended policy is that the research team will have exclusive use of the data for a period of 12 months from the end of the project, or until the data is published, if this is required alongside publications. Anonymised data will be provided and data will be made available upon application and the research team would control access in line with Northumbria University guidelines, however, data access will not reasonably be refused. There is no provision for public access to the protocol, statistical code and dataset, although reasonable requests will be accommodated in line with the intended use policy stated above.